CLINICAL TRIAL: NCT06947265
Title: Safety And Efficacy Of L-Arginine Monotherapy Versus Tadalafil Monotherapy Versus Their Combination In Men With Erectile Dysfunction; A Prospective Randomized Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Dogha, lecturer of urology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D 355
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Erectile Dysfunctions
Keywords: erectile dysfunction , L-arginine , elastography
MeSH Terms: conditions — Erectile Dysfunction | interventions — Arginine; Tadalafil

STUDY DESIGN:
Intervention Model Description: Group (1) was given daily 3 g(three divided doses) oral tablets of L-arginine for eight weeks.
  Group (2) was given daily 5 mg oral tablets of Tadalafil for eight weeks. Group (3) was given daily 3 g oral tablets of L-arginine and 5 mg oral tablets of Tadalafil for eight weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): was given daily 3 g(three divided doses) oral tablets of L-arginine for eight weeks
  Interventions: Drug: L-Arginine
- Group B (Experimental): was given daily 5 mg oral tablets of Tadalafil for eight weeks.
  Interventions: Drug: Tadalafil 5 mg
- Group C (Experimental): was given daily 3 g oral tablets of L-arginine and 5 mg oral tablets of Tadalafil for eight weeks.
  Interventions: Drug: L-Arginine; Drug: Tadalafil 5 mg

INTERVENTIONS:
Drug: L-Arginine — get 3 gm oral tablets of L-arginine
  Arms: Group A; Group C
Drug: Tadalafil 5 mg — get 5 mg oral tadalafil for 8 weeks
  Arms: Group B; Group C

SUMMARY:
Introduction Sexual dysfunctions are annoying health problems with the erectile problems forming the main part of them. Erectile dysfunction (ED) is defined as the persistent inability to obtain or maintain an erection that is sufficient to allow satisfactory sexual intercourse.[1] Aim of Work To evaluate the role of L-arginine monotherapy versus Tadalafil monotherapy versus their combination for the treatment of erectile dysfunction .

Patients and methods:

Inclusion criteria:

• Naive ( not previously treated) male patient with mild to moderate ED according to SHIM Questionnaire.

Exclusion criteria:

* Kidney disease or liver failure
* Coronary heart disease
* Peyronie's disease
* Neurological disease that may related to ED

DETAILED DESCRIPTION:
Safety And Efficacy Of L-Arginine Monotherapy Versus Tadalafil Monotherapy Versus Their Combination In Men With Erectile Dysfunction; A Prospective Randomized Study

Introduction Sexual dysfunctions are annoying health problems with the erectile problems forming the main part of them. Erectile dysfunction (ED) is defined as the persistent inability to obtain or maintain an erection that is sufficient to allow satisfactory sexual intercourse.[1] It is difficult to obtain accurate values for the true prevalence of erectile dysfunction, as many patients fail to seek any medical attention The best available data according to the Massachusetts Male Aging Study indicates that 52% of males between 40 and 70 years of age are affected with erectile problems, and about 70% of males are having some subjective issues with erections at the age of 70 years.[2] Erection is a neurovascular event in which a key mediator is nitric oxide (NO). It has been shown that there is reduced NO bioactivity in ED.[3] Oral phosphodiesterase-5 inhibitors (PDE-5 inhibitors), such as sildenafil and Tadalafil, are usually the first-line treatment of erectile dysfunction. They are effective in a wide range of etiologies including cardiovascular disease, diabetes, and hypogonadism. They act by decreasing the degradation of cyclic GMP via phosphodiesterase inhibition, which increases the relaxation of cavernosal smooth muscle and cavernosal arterial blood flow. It is important to note that PDE-5 inhibitors do not initiate the erectile response. Sexual stimulation is required to release nitric oxide from the vascular endothelium and penile nerve endings to commence the erectile process. PDE-5 inhibitors are highly effective and have an overall success rate of up to 76%.[4]

As L-arginine is a natural precursor of NO and its good availability is understood to have positive effect on NO production. Data regarding the pattern of use of L-arginine for sexual problems, which is considered one of the more widely used alternatives or adjuncts to regular drugs used in the patients of ED.[5] Aim of Work To evaluate the role of L-arginine monotherapy versus Tadalafil monotherapy versus their combination for the treatment of erectile dysfunction .

Patients and methods This clinical prospective study will be carried out on patients attending urology clinic in Fayoum University Hospital with ED

Sample size :

Inclusion criteria:

• Naive ( not previously treated) male patient with mild to moderate ED according to SHIM Questionnaire.

Exclusion criteria:

* Kidney disease or liver failure
* Coronary heart disease
* Peyronie's disease
* Neurological disease that may related to ED Patients were randomized equally categorized into three treatment groups. All the patients were blinded regarding the nature of the received medications.

Group (1) was given daily 3 g(three divided doses) oral tablets of L-arginine for eight weeks.

Group (2) was given daily 5 mg oral tablets of Tadalafil for eight weeks. Group (3) was given daily 3 g oral tablets of L-arginine and 5 mg oral tablets of Tadalafil for eight weeks.

Patients were advised to practice intercourse twice to three times weekly. They were assessed before and after eight weeks of treatment Pretreatment assessment

* History taking: including medical and surgical history.
* Sexual history: onset and duration of ED and Sexual health inventory for men (SHIM) to evaluate severity of ED.
* BMI
* General medical and local genital examinations.
* LABORATORY INVESTIGATIONS:

After 12 hours of fasting, venous blood samples were drawn from all included patients before and at the end of eight weeks of treatment for total serum testosterone assessments between 8.00 and 12.00 am.

• Penile ultrasonography: Shear Wave Elastography (SWE): is a current radiologic modality can measure biologic tissue elasticity and gives elastogram which superimposed on the B-mode ultrasound which expresses tissue stiffness in numbers(kpasc)

Follow up assessment:

* First follow up visit is scheduled after one week :to evaluate any adverse effect from the treatment
* 2nd follow up visit after 8 weeks : Reassessment to the SHIM questionnaire and serum testosterone and SWE.

Statistical analysis Data from the 3 groups will be collected, compared and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Naive ( not previously treated) male patient with mild to moderate ED according to SHIM Questionnaire.

Exclusion Criteria:

* ● Kidney disease or liver failure

  * Coronary heart disease
  * Peyronie's disease
  * Neurological disease that may related to ED

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only male
Enrollment: 180 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
SHIM questionnaire | 8 weeks of treatment
  The SHIM (Sexual Health Inventory for Men) questionnaire is a commonly used tool for assessing erectile dysfunction (ED) in men. It is a brief, self-administered questionnaire that typically consists of five questions, with answers scored on a scale to help determine the severity of erectile dysfunction. The SHIM is widely used in both clinical practice and research to assess sexual health and function.
  Here are the key elements of the SHIM:
  Frequency of sexual activity (often using a scale from "almost never or never" to "almost always or always").
  Confidence in maintaining an erection (again, on a similar scale). Ability to achieve an erection. Erection firmness (whether the erection is hard enough for penetration). Satisfaction with the firmness of the erection.
  The scores are typically aggregated into one overall score, and depending on the score, it classifies the degree of erectile dysfunction:
  25-22: No erectile dysfunction 21-17: Mild erectile dysfunction 16-12: Mild to mod

SECONDARY OUTCOMES:
testosterone level | 8 weeks of treatment
  androgenic hormone changes in response to treatment
Shear Wave Elastography | 8 weeks of treatment
  a current radiologic modality can measure biologic tissue elasticity and gives elastogram which superimposed on the B-mode ultrasound which expresses tissue stiffness in numbers(kpasc)

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mahmoud Dogha, Al Fayyum, Keman Fares, Egypt

IPD SHARING:
Plan to Share IPD: Undecided